CLINICAL TRIAL: NCT06083012
Title: Clinical and Healthcare Economic OutcoMes From ReAl-worlD Use in Europe of an AI Software During AF Ablation
Acronym: COMRADE-AI
Status: Active, not recruiting | Type: Observational
Sponsor: Volta Medical (Industry)
Collaborators: Fortrea (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIPL-01-004
Record Dates: First submitted 2023-10-09; First posted 2023-10-13 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation; Atrial Arrhythmia; Arrhythmias, Cardiac
Keywords: Artificial Intelligence; Cardiac ablation; Medical device; Software; Volta Medical; Atrial Arrhythmia; VX1; Volta AF-Xplorer; Volta AF-Xplorer II
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Cardiac mapping — All patients enrolled are treated for their atrial fibrillation/tachycardia via a catheter ablation procedure using VX1/Volta AF-Xplorer/Volta AF-Xplorer II software (used in accordance with its approved indication as per of its IFU) during the mapping phase to identify areas of interest specific to the patient.
  The ablation approach is free and chosen by the operator according to his standard practice. The two main phases of the ablation procedure are:
  * 3D mapping of the atria and location of areas of interest;
  * Catheter ablation at the operator's discretion.
  Other Names: Atrial fibrillation mapping; Ablation procedure

SUMMARY:
The goal of this Observational Prospective Multi-center Study is to observe the acute and long-term safety and performance outcomes after spatiotemporal dispersion-based AF/AT ablation utilizing the Volta Medical AI software in "real-life" clinical practice, without any imposed clinical workflow. Moreover, this study will allow to collect medico-economic data related to the tailored ablation strategy guided by the Volta Medical AI software.

DETAILED DESCRIPTION:
All patients enrolled are treated for atrial fibrillation/tachycardia via a catheter ablation procedure using Volta Medical AI software during the mapping phase to identify areas of interest specific to the patient. The ablation approach is free and chosen by the operator according to standard practice. Intraoperative and postoperative follow-up will be performed as in routine clinical practice during AF ablation procedures: hospitalization for ablation procedure and standard postoperative quarterly visits (at 3 months, at 6 months and/or 9 months as per the study investigator's Standard Of Care) then annual visits up to 24 months post-ablation. Adverse Events, recurrences of atrial arrhythmia and AF related symptoms (EHRA score) are collected from the patient's enrollment until the patient's study termination. A quality-of-life questionnaire related to general health (EQ-5D-3L) is collected during the preoperative visit and at least during annual follow-up visits. The patient's study-termination corresponds to the last annual visit at 24 months post-ablation index.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged 18 years or older.
2. Patient candidate for catheter ablation to treat paroxysmal or persistent atrial fibrillation, atrial tachycardia, de novo or after one or several previous ablation procedures, and for which the investigator considers using VX1 or Volta AF-Xplorer or Volta AF-Xplorer II.
3. Patient able and willing to provide written informed consent to participate in the study.
4. Only for France: Patient affiliated to the French social security system.

Exclusion Criteria:

1. Contraindication to AF/AT catheter ablation.
2. Patient who is or could potentially be pregnant.
3. Person deprived of liberty or under guardianship.
4. Person unable to undergo a medical monitoring for geographical, social or psychological reasons.
5. Patient's refusal to participate in the study.
6. Enrollment in an investigational study evaluating another device, biologic, or drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patient candidate eligible for catheter ablation to treat paroxysmal or persistent atrial fibrillation, atrial tachycardia, de novo or after one or several previous ablation procedures, and for which the investigator considers using VX1 or Volta AF-Xplorer or Volta AF-Xplorer II.
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2023-10-27 (Actual); Primary Completion 2027-04-27 (Estimated); Study Completion 2027-04-27 (Estimated)

PRIMARY OUTCOMES:
Freedom from clinically significant AF or atrial arrhythmia recurrence, after one or multiple ablation procedures, with or without antiarrhythmic drugs, stratified by type of clinical workflow. | [24 months]
VX1/Volta AF-Xplorer/Volta AF-Xplorer II-related Incident rate during ablation procedure. | [24months]
VX1/Volta AF-Xplorer/Volta AF-Xplorer II-related Adverse Event rate. | [24months]

SECONDARY OUTCOMES:
Progression of Quality-Of-Life score ("EQ-5D-3L") during the study (at inclusion, at quarterly visits, at 12 months and at 24 months). | Preoperative; [24months]
Progression of the AF related symptom score ("EHRA") during the study (at inclusion, at quarterly visits, at 12 months and at 24 months). | Preoperative; [24months]
Hospitalization rate during the post-ablation follow-up period. | [24months]
Serious Adverse Event rate during the post-ablation follow-up period. | [24months]
Average number of ablation procedures per patient up to 24 months follow-up. | [24months]
Average number of cardioversions per patient up to 24 months follow-up | [24months]
Progression of patient proportion under antiarrhythmic drugs and/or anticoagulant treatments during the study. | [24months]
Health economics analysis including QALY metric. | [24months]

CONTACTS AND LOCATIONS:
Overall Officials: Julien SEITZ, MD, Principal Investigator — Hôpital Saint Joseph Marseille
Locations (7):
- France (6):
  - Hôpital Saint-Joseph, Marseille
  - Hôpital Privé Jacques Cartier, Massy
  - Polyclinique Saint George, Nice
  - Centre Cardiologique du Nord, Saint-Denis
  - Clinique Rhéna, Strasbourg
  - Clinique Pasteur, Toulouse
- German Heart Center Munich, München, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seitz J, Bars C, Theodore G, Beurtheret S, Lellouche N, Bremondy M, Ferracci A, Faure J, Penaranda G, Yamazaki M, Avula UM, Curel L, Siame S, Berenfeld O, Pisapia A, Kalifa J. AF Ablation Guided by Spatiotemporal Electrogram Dispersion Without Pulmonary Vein Isolation: A Wholly Patient-Tailored Approach. J Am Coll Cardiol. 2017 Jan 24;69(3):303-321. doi: 10.1016/j.jacc.2016.10.065. PMID 28104073
- [Background] Seitz J, Durdez TM, Albenque JP, Pisapia A, Gitenay E, Durand C, Monteau J, Moubarak G, Theodore G, Lepillier A, Zhao A, Bremondy M, Maluski A, Cauchemez B, Combes S, Guyomar Y, Heuls S, Thomas O, Penaranda G, Siame S, Appetiti A, Milpied P, Bars C, Kalifa J. Artificial intelligence software standardizes electrogram-based ablation outcome for persistent atrial fibrillation. J Cardiovasc Electrophysiol. 2022 Nov;33(11):2250-2260. doi: 10.1111/jce.15657. Epub 2022 Sep 18. PMID 35989543
- [Background] Deisenhofer I. Electrogram-based AF ablation: finally, reproducibility! J Cardiovasc Electrophysiol. 2022 Nov;33(11):2261-2262. doi: 10.1111/jce.15660. Epub 2022 Sep 18. No abstract available. PMID 35989539